CLINICAL TRIAL: NCT04665882
Title: Intraoperative Nomogram to Predict Breast Cancer- Related Lymphedema Based in Artificial Intelligence Image Recognition: a Randomized Controlled Trial
Brief Title: Nomogram to Predict Breast Cancer Related Lymphedema
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wuhan University (Other)
Responsible Party: Principal Investigator, Gaosong Wu, Ph D, MD, Director, Wuhan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ZNJC201935
Record Dates: First submitted 2020-12-07; First posted 2020-12-14 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Breast Cancer; Axillary Lymph Node Dissection; Breast Cancer Related Lymphedema; Axillary Reverse Mapping
MeSH Terms: conditions — Breast Neoplasms; Breast Cancer Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Axillary surgery based on lymphedema prediction nomogram (Experimental): Based on the intraoperative lymphedema prediction nomogram, individualized treatment was recommended to breast cancer patients with different level of risk. For patients with low possibility of developing breast cancer related lymphedema, it was not necessary to preserve arm lymphatics. While the breast cancer patients who were performed mastectomy and ALND with 28 kg/m2 prepared to receive taxane-based chemotherapy, supraclavicular and infraclavicular radiotherapy, according to the established intraoperative nomogram, the proportion of the arm lymph flow above the axillary vein needed to exceed 52%. Otherwise, the arm lymphatics should be identified and preserved.
  Interventions: Procedure: Axillary surgery based on lymphedema prediction nomogram
- Standard axillary lymph node dissection (No Intervention): Standard axillary lymph node dissection was performed with complete resection of Berg's levels I and II.

INTERVENTIONS:
Procedure: Axillary surgery based on lymphedema prediction nomogram — Based on the intraoperative lymphedema prediction nomogram, individualized treatment was recommended to breast cancer patients with different level of risk. For patients with low possibility of developing breast cancer related lymphedema, it was not necessary to preserve arm lymphatics. While the breast cancer patients who were performed mastectomy and ALND with 28 kg/m2 prepared to receive taxane-based chemotherapy, supraclavicular and infraclavicular radiotherapy, according to the established intraoperative nomogram, the proportion of the arm lymph flow above the axillary vein needed to exceed 52%. Otherwise, the arm lymphatics should be identified and preserved.
  Arms: Axillary surgery based on lymphedema prediction nomogram

SUMMARY:
It has been hypothesized that damaged arm lymphatic drainage is associated with the arm lymphedema after axillary lymph node dissection (ALND). However, the majority of breast cancer patients with complete ALND has not suffered from arm lymphedema, which appears to be due to the residual arm lymph nodes that has not been removed in the axillary dissection. With the compensation of the residual arm lymph flow above the level of axillary vein, the arm lymphatic drainage could keep balance and remain normal function.

This arm lymphedema prediction model that included the protective factor, the proportion of arm lymph flow above the level of axillary vein, allows intraoperative intervention to be performed for the high-risk group. The arm lymphatics of these distinguished patients would be preserved to eliminate the occurrence of arm lymphedema in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older with T1-3 invasive breast cancer;
* Clinically node-positive breast cancer, defined as positive on preoperative axillary palpation, ultrasound examination, and computed tomography scan with contrast;
* Patients who underwent mastectomy with a positive sentinel lymph node (SLN);
* Patients who underwent breast-conserving surgery containing more than two positive SLNs.

Exclusion Criteria:

* Neoadjuvant chemotherapy;
* Previous history of breast cancer.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2020-12-11 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of arm lymphedema | Up to 5 years
  A difference in volume between the arms < 10% was defined as lymphedema
Rate of locoregional recurrence | Up to 5 years
  Locoregional recurrence included local recurrence and regional recurrence. Local recurrence was defined as chest wall recurrence of breast cancer, and regional recurrence was defined as the axilla recurrence of breast cancer
Rate of distant metastasis | Up to 5 years
  Cancer cells from breast metastasized to other organs.

CONTACTS AND LOCATIONS:
Overall Officials: Gaosong Wu, Ph.D., Principal Investigator — Wuhan University
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided